CLINICAL TRIAL: NCT06387238
Title: Exploration of the Value of PSMA PET/CT in Dynamic Monitoring of the Efficacy of Novel Endocrine Therapy in Patients With Metastatic Hormone Sensitive Prostate Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PSMA-mHSPC
Record Dates: First submitted 2024-03-27; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Prostate Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: Patients With Metastatic Hormone Sensitive Prostate Cancer, will receive pre-therapeutic PSMA PET/CT and post-therapeutic PSMA PET/CT after three-month novel endocrine therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mHSPC-PSMA (Experimental): Patients with mHSPC who will receive pre-therapeutic PSMA PET/CT and post-therapeutic PSMA PET/CT after three-month novel endocrine therapy.
  Interventions: Diagnostic Test: PSMA PET/CT

INTERVENTIONS:
Diagnostic Test: PSMA PET/CT — pre-therapeutic PSMA PET/CT and post-therapeutic PSMA PET/CT after three-month novel endocrine therapy.

SUMMARY:
1. Based on the treatment response and prognosis of mHSPC patients with novel endocrine therapy, a PSMA PET whole-body tumor burden classification was constructed to guide treatment and evaluate prognosis.
2. Based on the treatment response and prognosis of mHSPC patients with novel endocrine therapy, a multivariable model will be constructed using quantitative parameters of PSMA PET/CT imaging, pre-treatment gene status, PSA, GS/ISUP and other clinical pathological parameters to further achieve accurate patient classification, guide treatment, and evaluate prognosis.

DETAILED DESCRIPTION:
1. Construction of PSMA PET whole-body tumor burden classification:

1. Assessment of whole-body tumor burden on PSMA PET/CT images of mHSPC patients before new endocrine therapy.
2. PSMA PET/CT imaging evaluation of treatment response of the first three months after start of new endocrine therapy.
3. Based on the response results, the optimal threshold for whole-body tumor burden is obtained through ROC curve analysis, and a preliminary classification of whole-body tumor burden is obtained.

Verification 1: Follow up preliminary verification/improvement of this subtype Verification 2: External verification, reverifying the predictive performance of typing through the verification cohort.

2. Construction of multivariable predictive model for mHSPC patients with novel endocrine therapy:

1. Molecular imaging parameter measurement and collection of PSMA PET/CT images of mHSPC patients of 3 months after the start of new endocrine therapy.
2. Complete pre-treatment genetic testing, dynamic evaluation of serum PSA before and after treatment, and collection of clinical and pathological information.
3. Based on follow-up results, construct a multi factor model, screen significant factors, and achieve a predictive model for novel endocrine therapy in mHSPC patients Verification: External verification, verifying the predictive performance of the model through the verification cohort.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients confirmed to have metastasis by PSMA PET/CT before new endocrine therapy.

  * Those who have not undergone androgen deprivation treatment in the past, or have currently received androgen deprivation treatment for no more than 120 days without progress, or have received androgen deprivation treatment in the past (treatment time less than 24 months and no progress within 12 months after completion).

    * Patients with KPS score ≥ 50 (ECOG/WHO equivalent).

      * Patient age>18 years old.

Exclusion Criteria:

Patients who cannot understand and voluntarily participate in this trial, donnot sign an informed consent form, and aren't able to cooperate independently in completing the examination.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
rPFS | From date of enrollment treatment until the date of first documented progression confirmed by radiological examinations or date of death from any cause, whichever came first, assessed up to 12 months.
  radiological progression free survival

SECONDARY OUTCOMES:
PSA-PFS | From date of enrollment treatment until the date of first documented progression confirmed by blood PSA tests or date of death from any cause, whichever came first, assessed up to 12 months.
  PSA progression free survival
OS | From date of enrollment treatment until the date of death from any cause, assessed up to 12 months.
  overall survival

IPD SHARING:
Plan to Share IPD: No